CLINICAL TRIAL: NCT05320367
Title: A Randomized, Triple Blinded Cross-over Placebo Controlled Study of Effects of Inhaled Cannabidiol in Healthy Occasional Cannabis Users
Brief Title: A Study of Inhaled Cannabidiol in Healthy Occasional Cannabis Users
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21.361
Record Dates: First submitted 2022-03-20; First posted 2022-04-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: In this crossover design, participants will be administered both dosages of CBD and placebo during participation in the study. Participant will be randomly assigned to one of ten pre-determined sequences with a CBD or placebo product at 5 dosages (0 mg, 5 mg, 20 mg, 50 mg and 100 mg). Participants will be randomized based on a completely balanced 5 by 5 latin square
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CBD (Group 1) (Experimental): Group will receive four CBD doses (5 mg, 20 mg, 50 mg and 100 mg), and placebo (0 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence
  Interventions: Drug: Cannabis, placebo
- CBD (Group 2) (Experimental): Group will receive four CBD doses (5 mg, 20 mg, 50 mg and 100 mg), and placebo (0 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence
  Interventions: Drug: Cannabis, placebo
- CBD (Group 3) (Experimental): Group will receive four CBD doses (5 mg, 20 mg, 50 mg and 100 mg), and placebo (0 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: Cannabis, placebo
- CBD (Group 4) (Experimental): Group will receive four CBD doses (5 mg, 20 mg, 50 mg and 100 mg), and placebo (0 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: Cannabis, placebo
- CBD (Group 5) (Experimental): Group will receive four CBD doses (5 mg, 20 mg, 50 mg and 100 mg), and placebo (0 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: Cannabis, placebo

INTERVENTIONS:
Drug: Cannabis, placebo — Eligible participant will be randomize 1:1:1:1:1 to receive placebo, CBD (5mg, 20mg, 50mg and 100mg). Only one research product will be inhaled for each visit. The sequence will depend on the assigned randomization group.

SUMMARY:
The purposes of this study are 1) to determine if the administration of different low doses of CBD (5 mg, 20 mg, 50 mg and 100 mg) result in detectable subjective pleasant drug effect compared to placebo and 2) to qualitatively explore whether low dose CBD is associated with effects that are not detected with the available research tools.

DETAILED DESCRIPTION:
Cannabis contains over 100 cannabinoids, the two most prominent being Δ-9-tetrahydrocannabinol (THC) and cannabidiol (CBD). A growing body of evidence exists surrounding the effects of both THC and CBD, however, less is known about the specific effects of CBD concentrations alone. Most existing data regarding the effects of CBD come from studies where this compound is administered in high doses in a therapeutic context, and where the subject can be administered either CBD, THC or both together. These contexts are not representative of the current use by many consumers. Indeed, several available products contain CBD at much lower doses. The overall objective of this study is to evaluate the acute behavioral and biological effects of low doses of CBD (between 5-100mg) and placebo in occasional cannabis users. Potential outcomes not detected with usual assessment tools designed to evaluate THC-induced effects will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Between 21 and 49 years of age, inclusively;
2. Have used cannabis at least once in lifetime AND have used cannabis three days or less in the 28 days prior to enrollment;
3. Be able to provide a signed informed consent;
4. Willing to comply with study procedures and requirements as per protocol, including to abstain from using other cannabis products or any drugs (except alcohol or nicotine) 7 days prior to study visits;
5. Have a forced expiratory volume in first second (FEV) sup 90 %;
6. Able to communicate and understand English or French language;
7. For female participants:

   a. Without childbearing potential, defined as: i. postmenopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age); or ii. Documented surgically sterilized (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or

   b. With childbearing potential: i. Must have negative pregnancy test result at screening and at subsequent visits.

ii. AND have no pregnancy plan while on the trial iii. AND must agree to use a medically accepted method of birth control throughout the study.

Exclusion Criteria:

1. Any disabling medical conditions, as assessed by medical history, physical exam, vital signs and/or laboratory assessments that, in the opinion of the study physician, precludes safe participation in the study or the ability to provide fully informed consent;
2. Severe psychiatric condition (e.g. history of schizophrenia, schizoaffective disorder or bipolar disorder; current acute psychosis, mania or current suicidality, acute depression or anxiety disorder based on the Mini International Neuropsychiatric Interview);
3. Any other disabling, unstable, or acute mental condition that, in the opinion of the study physician, precludes safe participation in the study or ability to provide informed consent;
4. Known chronic liver disease or aspartate transaminase/alanine transaminase (AST/ALT) two times higher than upper limit of normal values at screening visit;
5. Blood pressure higher than 130/80 mmHg;
6. Kidney disorders;
7. Bleeding disorders;
8. Current moderate or severe DSM-5 (The Diagnostic and Statistical Manual of Mental Disorders) substance use disorder (except nicotine) according to the Structured Clinical Interview for DSM-V ;
9. Currently pregnant,breastfeeding or planning to become pregnant either at screening or while enrolled in the study;
10. Pending legal action or other reason that, in the opinion of the study physician, might prevent study completion;
11. Use of medication within 7 days of experimental sessions, which, in the opinion of the investigator, may interact with cannabis;
12. Participation in clinical studies or undergoing other investigational procedures involving cannabis or cannabinoids administration within 30 days prior to randomization;
13. Resting heart rate over 100 beats per minute;
14. Current body mass index (BMI) over 29.9 kg/m2;
15. Any clinically significant electrocardiogram abnormalities at screening visit.

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pleasant drug effect | T1(10 minutes after inhalation)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).
Pleasant drug effect | T2 (80 minutes after inhalation)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).
Pleasant drug effect | T3 (140 minutes after inhalation)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).

SECONDARY OUTCOMES:
Drug Effects associated with cannabis administration | T1 (10 minutes after inhalation)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis administration and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Drug Effects associated with cannabis administration | T2 (80 minutes after inhalation)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis administration and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Drug Effects associated with cannabis administration | T3 (140 minutes after inhalation)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis administration and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Change in dissociation | Baseline and after inhalation at (10 minutes, 80 minutes)
  Dissociation will be assessed using the Clinician Administered Dissociative States Scale (CADSS) administered at Baseline (T0) and following administration of the study product (T1- 10 minutes, T2-60 minutes) at each study visit. The CADSS, a 28-items validated instrument, includes 5 observer items and 23 participant self-report items rated on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). Minimum score :0 not at all; Maximum score 72 extremely dissociate.
Cannabis-Specific Subjective Effects | T3 (140 minutes after inhalation)
  Subjective effects of cannabis will be assessed using both the positive and negative subscales of the Cannabis Experience Questionnaire administered following administration study product. Each item is rated on a 5-point scale, ranging from 1 (not at all) to 5 (severely).The positive subscale includes16 items related to euphoric experiences (maximum 90 and minimum 16). The negative subscale includes 25 items related to paranoid-dysphoric experiences (Maximum 125 and minimum 25).
Change in Affect | Baseline and after inhalation at (10 minutes, 80 minutes, 140 minutes)
  Affect will be measured using the Positive and Negative Affect Schedule administered at Baseline (T0) and following administration of the study product at each study visit. The Positive and Negative Affect Schedule is a 20-item validated questionnaire divided into subscales of positive (10 items) and negative affect (10 items). Each item is rated on a 5-point scale ranging from 1 (not at all) to 5 (extremely). For each subscale minimum is 10 and maximum 50.
Change in Anxiety Symptoms | Baseline and after inhalation at (10 minutes, 80 minutes and 140 minutes)
  Symptoms of anxiety will be assessed using the States-Trait-Anxiety-Inventory, a 20-item validated self-report scale that measures the severity of anxiety in adults.. Each symptom is rated on a 4-point scale ranging from 1 (not at all) to 4 (very much).
Change in Safety | Baseline and after inhalation at (10 minutes, 80 minutes, 140 minutes)
  Adverse events will be collected prior to administration of the study product (T0) and following administration of the study product (T1, T2 and T3)
Change on cognition | Baseline and after inhalation at T2 (80 minutes).
  The Cambridge Neuropsychological Test Automated Battery tests will be used for the rapid assessment of multiple cognitive components.
Visit Intoxication Assessment | End of the visit, approximatively 180 minutes after inhalation
  Signs of intoxication will be assess using the modified Standardized Field Sobriety Test.

OTHER OUTCOMES:
Change in plasma concentration of CBD | Baseline and after inhalation at ( 5 minutes, 15 minutes, 80 minutes, 110 minutes, 140 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after inhalation.
Change in plasma concentration of 7-Hydroxycannabidiol | Baseline and after inhalation at ( 5 minutes, 15 minutes, 80 minutes, 110 minutes, 140 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after inhalation.
Change in plasma concentration of 7-Carboxy-Cannabidiol | Baseline and after inhalation at ( 5 minutes, 15 minutes, 80 minutes, 110 minutes, 140 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after inhalation.
Change in plasma concentration of Anandamide | Baseline and after inhalation at ( 5 minutes, 15 minutes, 80 minutes, 110 minutes, 140 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD,MS, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)

IPD SHARING:
Plan to Share IPD: No